CLINICAL TRIAL: NCT00590096
Title: I-123-MIBG for Imaging of Neuroblastoma and Pheochromocytoma
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: University of Cincinnati (Other)
Responsible Party: Michael J. Gelfand M.D., Cincinnati Children's Hospital
Other Study IDs: CCHMC# 88-12-2
Record Dates: First submitted 2007-12-27; First posted 2008-01-10 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2007-01

CONDITIONS: Neuroblastoma; Pheochromocytoma
Keywords: Neuroblastoma; Pheochromocytoma; MIBG
MeSH Terms: conditions — Neuroblastoma; Pheochromocytoma

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

SUMMARY:
I-123-MIBG is used to image patients with neuroblastoma, pheochromocytoma and other neural crest tumors

DETAILED DESCRIPTION:
Entry criteria--Histologically documented neuroblastoma or pheochromocytoma or strong suspicion of neuroblastoma or pheochromocytoma.

Exclusion criteria--Pregnancy Randomization--None Procedure--Patients will receive a dose of I-123-MIBG by intravenous injection. Images will obtained at 18-24 hours after administration of the drug and at 42-48 hours as needed. SSKI will be used to block thyroid uptake of free I-123-iodide

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven neuroblastoma or pheochromocytoma or strong suspicion of neuroblastoma or pheochromocytoma

Exclusion Criteria:

* Pregnancy

Min Age: 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with histologically proven neuroblastoma or pheochromocytoma or strong suspicion of neuroblastoma or pheochromocytoma
Sampling Method: Non-Probability Sample
Enrollment: 1380 (Actual)
Dates: Start 1991-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Gelfand, M.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati

REFERENCES:
- [Background] Chan EL, Harris RE, Emery KH, Gelfand MJ, Collins MH, Gruppo RA. Favorable histology, MYCN-amplified 4S neonatal neuroblastoma. Pediatr Blood Cancer. 2007 Apr;48(4):479-82. doi: 10.1002/pbc.20705. PMID 16333837
- [Background] Gelfand MJ. 123I-MIBG uptake in the neck and shoulders of a neuroblastoma patient: damage to sympathetic innervation blocks uptake in brown adipose tissue. Pediatr Radiol. 2004 Jul;34(7):577-9. doi: 10.1007/s00247-003-1136-x. Epub 2004 Mar 3. PMID 15205842
- [Background] Gelfand MJ. Meta-iodobenzylguanidine in children. Semin Nucl Med. 1993 Jul;23(3):231-42. doi: 10.1016/s0001-2998(05)80104-7. PMID 8378796
- [Result] Gelfand MJ, Elgazzar AH, Kriss VM, Masters PR, Golsch GJ. Iodine-123-MIBG SPECT versus planar imaging in children with neural crest tumors. J Nucl Med. 1994 Nov;35(11):1753-7. PMID 7965151
- [Result] Paltiel HJ, Gelfand MJ, Elgazzar AH, Washburn LC, Harris RE, Masters PR, Golsch GJ. Neural crest tumors: I-123 MIBG imaging in children. Radiology. 1994 Jan;190(1):117-21. doi: 10.1148/radiology.190.1.8259387.
- [Result] Englaro EE, Gelfand MJ, Harris RE, Smith HS. I-131 MIBG imaging after bone marrow transplantation for neuroblastoma. Radiology. 1992 Feb;182(2):515-20. doi: 10.1148/radiology.182.2.1732972.
- [Result] Elgazzar AH, Gelfand MJ, Washburn LC, Clark J, Nagaraj N, Cummings D, Hughes J, Maxon HR 3rd. I-123 MIBG scintigraphy in adults. A report of clinical experience. Clin Nucl Med. 1995 Feb;20(2):147-52. doi: 10.1097/00003072-199502000-00011. PMID 7720307